CLINICAL TRIAL: NCT05291247
Title: Physician-Initiated PMCF Trial Investigating Shockwave Intravascular Lithotripsy and a Drug Eluting Vascular Stent System Deployment for Heavily Calcified Femoropopliteal Disease
Brief Title: Shockwave IVL + DES
Acronym: Shockwave DES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Sabrina Overhagen (Other)
Responsible Party: Sponsor-Investigator, Dr. Sabrina Overhagen, Director, FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Other Study IDs: FCRE-210505
Record Dates: First submitted 2021-11-21; First posted 2022-03-22 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Arterial Disease; Superficial Femoral Artery Stenosis; Calcifications Vascular
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heavily calcified femoropopliteal disease: * Subject must be between 21 and 85 years old
  * Clinical diagnosis of symptomatic peripheral artery disease, defined by Rutherford Becker Classification score 3-5
  * Willing to comply with the specified follow-up evaluation
  * Written informed consent prior to any study procedures
  Interventions: Device: Peripheral lithotripsy system (Shockwave Medical)

INTERVENTIONS:
Device: Peripheral lithotripsy system (Shockwave Medical) — The combination of Shockwave Intravascular Lithotripsy and a polymer coated Drug Eluting Stent device for calcified femoropopliteal disease.

SUMMARY:
The objective of this clinical investigation is to evaluate, in a controlled setting, the 12 months safety and efficacy of the combination of Shockwave Intravascular Lithotripsy and a polymer coated Drug Eluting Stent device, for PACSS 3 and PACSS 4 calcified femoropopliteal disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 21 and 85 years old
* Clinical diagnosis of symptomatic peripheral artery disease, defined by Rutherford Becker Classification score 3-5
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures
* Stenotic, restenotic after PTA or occlusive lesion(s) located in the native Superficial Femoral Artery (SFA) and/or proximal Popliteal Artery (PPA):

  1. Degree of stenosis ≥ 70% by visual agiographic assessment
  2. Vessel diameter ≥ 4 and ≥ 6 mm
  3. Total lesion length (or series of lesions) ≥ 30 mm and 210 mm (Note: Lesion segment(s) must be filly covered with one or two overlapping DES stent (s) be fully covered with one or two overlapping DES stent(s)
  4. Target lesion located at least three centimeters above the inferior edge of the femur
* Severity of calcification PACSS 3-4
* Patent infrapopliteal and popliteal artery; i.e. single vessel runoff or better with at least one of three vessels patent (>50% stenosis) to the ankle or foot with no planned intervention.
* Study entry after successful target lesion crossing of the guidewire (guidewire located intraluminally or subintimally); Both crossing devices as well as retrograde recanalization can be used.
* Non-target lesion interventions to restore adequate blood flow, in the same index procedure are allowed. This intervention must be prior to the treatment of the study lesion and should be completed successfully.

Exclusion Criteria:

* Not treated ipsilateral significant (>50%) stenosis of the iliac arteries
* Non severely calcified disease (absence of calcification, PACSS 1, PACSS 2)
* Significant (>50%) stenosis of all infrapopliteal arteries, no patent artery to the foot
* Angiographic evidence of thrombus within the target vessel
* Thrombolysis within 72 hours prior to the index procedure
* Previously stented target lesion / vessel
* Subjects who have undergone prior surgery of the target lesion SFA/PPA to treat atherosclerotic disease
* Bypass Anastomosis stenosis
* Concomitant hepatic insufficiency, thrombophlebitis, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Recent MI or stroke <30 days prior to the index procedure
* Life expectancy less than 24 months
* Known or suspected active infection at the time of the index procedure
* Known or suspected major allergies or contraindications to aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, or contrast agent
* Any significant medical condition which, in the investigator's opinion, may interfere with the subject's optimalparticipation in the study
* The subject is currently participating in another drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
* Female subjects pregnant, breastfeeding, of childbearing potential who are planning to become pregnant in the next 5 years.
* End-stage-renal disease
* Presence of Severe Ischemic Ulcers or frank gangrene (Rutherford class 6).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population for this study are patients with a diminished blood flow in their heavily calcified femoropopliteal lesions, who need a reintervention.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 12 months
  Defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.4) and without Target Lesion Revascularization (TLR)
Procedural success: | 30 days post procedure
  Defined as technical success and completion of the procedure without complications , meaning successful treatment of the vessels (technical success) in the absence of:
  * vessel rupture or perforation that require an intervention
  * need for emergency surgical revascularization of target limb
  * symptomatic thrombus or distal emboli that require surgical, mechanical, or pharmacologic means to improve flow and extend hospitalization
  * unplanned above the ankle amputation
  * major adverse cardiovascular events (defined as composite of total death, myocardial infarction, coronary revascularization and stroke).

SECONDARY OUTCOMES:
Primary Patency | 6 months
  Defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50 systolic velocity ratio no greater than 2,4) and without Target Lesion Revascularization (TLR)
Target Lesion Revascularization (TLR) | 6- and 12-months
  Defined as the need for target lesion revascularization after index procedure.
Secondary Patency Rate | 6- and 12-months
  Defined as restored flow in the treated segment after occlusion or restenosis.
Amputation-free Survival rate | 6- and 12-months
  Defined as the time until a major amputation of the index limb and/or death of any cause, whichever occurred first.
Major Amputation Rate | 6- and 12-months
  Defined as any aboveankle amputation.
Clinical Success | 6- and 12-months
  Defined as an improvement of the Rutherford Becker Classification of one class or more, as compared to the preprocedure Rutherford Becker Classification.
Absence of Major Adverse Events (MAE) | 6- and 12-months
  Acute Coronary Syndrome, Stroke, Death, Major Amputation or TLR.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Stavroulakis, MD, Principal Investigator — Vascular Department, LMU Munich
Locations (6):
- Germany (6):
  - Klinikum Hochsauerland, Arnsberg
  - University Hospital Essen, Essen
  - University Hospital Eppendorf, Hamburg
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad
  - St. Marien Hospital, Lünen
  - University Hospital LMU Munich, Munich

IPD SHARING:
Plan to Share IPD: No